CLINICAL TRIAL: NCT01819571
Title: Pulse Pressure Variation for Prediction of Fluid Responsiveness in Coronary Artery Disease Patients With Diastolic Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1-2011-0056
Record Dates: First submitted 2013-03-14; First posted 2013-03-27 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Fluid Responsiveness Predictability
Keywords: pulse pressure variation; fluid responsiveness; diastolic dysfunction
MeSH Terms: interventions — HES 130-0.4

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal diastolic function group (Experimental)
  Interventions: Drug: Fluid loading (Voluven)
- Diastolic dysfunction group (Active Comparator)
  Interventions: Drug: Fluid loading (Voluven)

INTERVENTIONS:
Drug: Fluid loading (Voluven) — HES 130/0.4 (VoluvenⓇ, Fresenius Kabi, Graz, Austria) 8ml / kg loading during 15 minutes after induction of anesthesia on both groups
  Other Names: Fluid loading

SUMMARY:
The investigators hypothesized that predictability of pulse pressure variation (PPV) on fluid responsiveness would be reduced in patients with coronary disease who have diastolic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 20 years
* scheduled for elective coronary artery bypass grafting
* normal diastolic function (E/E' < 8) or diastolic dysfunction (E/E' >15) according to preoperative Echocardiographic evaluation

Exclusion Criteria:

* arrythmia,
* reduced left ventricular function (ejection fraction < 40%)
* valvular heart disease requiring concomitant surgical correction
* pulmonary hypertension (mean pulmonary arterial pressure ≥30 mm Hg)
* peripheral arterial occlusive disease, pulmonary disease (asthma, chronic obstructive pulmonary disease, and lung resection)
* end-stage renal disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
predictability of pulse pressure variation (PPV) on fluid responsiveness in patients with coronary disease who have normal diastolic function and diastolic dysfunction. | 10 minutes after fluid replacement
  After induction of anesthesia and applying mechanical ventilation, hemodynamic parameters (including PPV measured by Philips IntelliVue MP 70®) were recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Department of anesthesiology and pain medicine, Seoul, Seoul, South Korea